CLINICAL TRIAL: NCT02322775
Title: A Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled, Phase 3 Study to Evaluate the Efficacy and Safety of Benralizumab in Adult Patients With Mild to Moderate Persistent Asthma.
Brief Title: Study to Evaluate the Efficacy and Safety of Benralizumab in Adult Patients With Mild to Moderate Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D3250C00032; 2014-004427-40 (EudraCT Number)
Record Dates: First submitted 2014-12-19; First posted 2014-12-23 (Estimated); Results first posted 2017-02-14 (Actual); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: Asthma
Keywords: Asthma, Bronchial Diseases, Respiratory Tract Diseases, Lung Diseases, Obstructive Lung Diseases,
MeSH Terms: conditions — Asthma; Bronchial Diseases; Respiratory Tract Diseases; Lung Diseases; Lung Diseases, Obstructive | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Benralizumab administered subcutaneously every 4 weeks
  Interventions: Biological: Benralizumab
- Arm B (Experimental): Placebo administered subcutaneously every 4 weeks
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Benralizumab — Benralizumab administered subcutaneously every 4 weeks
  Arms: Arm A
Biological: Placebo — Placebo administered subcutaneously every 4 weeks
  Arms: Arm B

SUMMARY:
The purpose of this trial is to confirm the safety and clinical benefit of benralizumab administration in asthma patients with mild to moderate persistent asthma in order to gain an understanding of the benefit/risk of benralizumab across the spectrum of asthma disease.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent for study participation must be obtained prior to any study related procedures being performed and according to international guidelines and/or applicable European Union (EU) guidelines.

* Female and male aged 18 to 75 years, inclusively, at the time of Visit 1.
* Weight of ≥40 kg.
* Evidence of asthma as documented by post-bronchodilator (post-BD) reversibility in FEV1 of ≥ 12% demonstrated at Visit 2.
* Documented use of 1 of the following types of asthma therapy at time of informed consent: Low- to medium-dose ICS (ie, 100 to 500 μg fluticasone dry powder formulation equivalents total daily dose) with or without other controller medications, eg, an LTRA and/or theophylline or Low-dose ICS/LABA fixed combination therapy (eg, the lowest regular maintenance dose approved in the local country will meet this criterion)
* Morning pre-bronchodilator (pre-BD) FEV1 of > 50% to ≤ 90% predicted at Visit 2.

Exclusion Criteria:

* Clinically important pulmonary disease other than asthma (eg, active lung infection, COPD, bronchiectasis, pulmonary fibrosis, cystic fibrosis, hypoventilation syndrome associated with obesity, lung cancer, alpha 1 anti-trypsin deficiency, and primary ciliary dyskinesia) or ever been diagnosed with pulmonary or systemic disease, other than asthma, that are associated with elevated peripheral eosinophil counts (eg, allergic bronchopulmonary aspergillosis/mycosis, Churg-Strauss syndrome, hypereosinophilic syndrome).
* Any disorder, including, but not limited to, cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematological, psychiatric, or major physical impairment that is not stable in the opinion of the Investigator and could:
* Affect the safety of the patient throughout the study
* nfluence the findings of the studies or their interpretations,- Impede the patient's ability to complete the entire duration of study.
* Known history of allergy or reaction to the investigational product formulation.
* History of anaphylaxis to any biologic therapy.- History of Guillain-Barré syndrome.
* A helminth parasitic infection diagnosed within 24 weeks prior to the date informed consent is obtained that has not been treated with, or has failed to respond to standard of care therapy.- Acute upper or lower respiratory infections requiring antibiotics or antiviral medication within 30 days prior to the date informed consent is obtained or during the screening/run-in period.
* Any clinically significant abnormal findings in physical examination, vital signs, hematology, clinical chemistry, or urinalysis during screening period, which in the opinion of the Investigator, may put the patient at risk because of his/her participation in the study, or may influence the results of the study, or the patient's ability to complete entire duration of the study.
* Positive hepatitis B surface antigen, or hepatitis C virus antibody serology, or a positive medical history for hepatitis B or C. Patients with a history of hepatitis B vaccination without history of hepatitis B are allowed to enroll.
* A history of known immunodeficiency disorder including a positive human immunodeficiency virus (HIV) test.
* History of cancer:
* Patients who have had basal cell carcinoma, localized squamous cell carcinoma of the skin or in situ carcinoma of the cervix are eligible provided that the patient is in remission and curative therapy was completed at least 12 months prior to the date informed consent was obtained.
* Patients who have had other malignancies are eligible provided that the patient is in remission and curative therapy was completed at least 5 years prior to the date informed consent was obtained

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2015-02-02 (Actual); Primary Completion 2015-10-07 (Actual); Study Completion 2015-10-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary T. Ferguson, M.D.,P.C., Principal Investigator — Pulmonary Research Institute of Southeast Michigan
Locations (52):
- United States (17):
  - Research Site, Los Angeles, California
  - Research Site, Rolling Hills Estates, California
  - Research Site, Clearwater, Florida
  - Research Site, Orlando, Florida
  - Research Site, Blue Island, Illinois
  - Research Site, Skillman, New Jersey
  - Research Site, Charlotte, North Carolina
  - Research Site, Monroe, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Grove City, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Spartanburg, South Carolina
  - Research Site, El Paso, Texas
  - Research Site, San Antonio, Texas
- Canada (9):
  - Research Site, Vancouver, British Columbia
  - Research Site, Ajax, Ontario
  - Research Site, Burlington, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Québec, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Trois-Rivières, Quebec
- Germany (6):
  - Research Site, Bamberg
  - Research Site, Berlin
  - Research Site, Frankfurt
  - Research Site, Frankfurt am Main
  - Research Site, Hanover
  - Research Site, Neu-Isenburg
- Hungary (5):
  - Research Site, Balassagyarmat
  - Research Site, Komárom
  - Research Site, Miskolc
  - Research Site, Pécs
  - Research Site, Százhalombatta
- Poland (7):
  - Research Site, Katowice
  - Research Site, Mrągowo
  - Research Site, Ostrów Wielkopolski
  - Research Site, Pabianice
  - Research Site, Poznan
  - Research Site, Tarnów
  - Research Site, Wroclaw
- Slovakia (8):
  - Research Site, Bratislava
  - Research Site, Humenné
  - Research Site, Košice
  - Research Site, Levice
  - Research Site, Poprad
  - Research Site, Prešov
  - Research Site, Vráble
  - Research Site, Žilina

REFERENCES:
- [Background] Ferguson GT, FitzGerald JM, Bleecker ER, Laviolette M, Bernstein D, LaForce C, Mansfield L, Barker P, Wu Y, Jison M, Goldman M; BISE Study Investigators. Benralizumab for patients with mild to moderate, persistent asthma (BISE): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Respir Med. 2017 Jul;5(7):568-576. doi: 10.1016/S2213-2600(17)30190-X. Epub 2017 May 22. PMID 28545978
- See also: CSP redacted — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3365&filename=ClinicalStudyProtocol_BISE_redacted.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After enrollment, eligible patients entered a 2- to 4-week screening/run-in period and were converted to budesonide dry powder inhaler twice daily for the duration of the study.
  Patients who continued to meet eligibility criteria at the end of the run-in period entered a 12 weeks double-blind treatment period followed by two follow-up visits.
Pre-assignment Details: Eligible adult patients were stratified by baseline blood eosinophil count (<300 cells/μL or ≥300 cells/μL) and by region (USA versus Rest of the World per the IVRS). Patients were then randomized to either benralizumab 30 mg Q4W or placebo in a 1:1 ratio.
Groups:
- Benralizumab 30 mg Q4W: Benralizumab administered subcutaneously every 4 weeks
Period: Overall Study
Arm/Group | Benralizumab 30 mg Q4W | Placebo
Started | 106 | 105
Completed | 101 | 99
Not Completed | 5 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 3 | 4
Not completed — Not willing to perform all FU visits | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Benralizumab 30 mg Q4W | Placebo | Total
Number analyzed (Participants) | 106 | 105 | 211
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.3 (14.40) | 51.1 (12.60) | 49.7 (13.58)
Age, Customized [Number; unit: Participants]
  >=18-<50 years | 49 | 44 | 93
  >=50-<65 years | 43 | 46 | 89
  >=65-<=75 years | 14 | 15 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 67 | 129
  Male | 44 | 38 | 82
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 0 | 1
  Black or African American | 7 | 4 | 11
  White | 98 | 99 | 197
  Other | 0 | 2 | 2
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 100 | 102 | 202

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Pre-bronchodilator Forced Expiratory Volume in 1 Second (FEV1) (L) at Week 12
Description: The FEV1 (L) change from baseline are compared between benralizumab 30 mg Q4W and placebo by using the mixed-effect repeated measures (MMRM) analysis with baseline blood eosinophil count (≥300 cells/μL or <300 cells/μL), protocol specified visit (Week 4, Week 8, Week 12), region (Europe or North America) and treatment*visit interaction as fixed effects and baseline pre-bronchodilator FEV1 (L) as a covariate.
  Changes at Week 12 were calculated based on patients with both baseline and Week 12.
Time Frame: Baseline, Week 4, Week 8 and Week 12
Population: The Full Analysis Set comprised all patients randomised and receiving any investigational product (IP), irrespective of their protocol adherence and continued participation in the study.
Measure: Mean (Standard Deviation); unit: Litre
Arm/Group | Benralizumab 30 mg Q4W | Placebo
Number analyzed (Participants) | 106 | 105
Litre
  Baseline | 2.248 (0.6062) | 2.246 (0.7677)
  Week 12 | 2.310 (0.6702) | 2.261 (0.7959)
  Change from baseline at Week 12 | 0.057 (0.2734) | -0.016 (0.2350)
Statistical Analysis 1: Comparison: Benralizumab 30 mg Q4W vs Placebo; The null hypothesis was: H0: Change from baseline in pre-bronchodilator FEV1 (L) at Week 12 (benralizumab vs placebo)=0; Test type: Superiority or Other; p = 0.040, Mixed Models Analysis — Hypothesis testing were reported using 2-sided 5% level tests with nominal p-values (i.e., not adjusted for multiplicity); Difference of Least Square Means = 0.08, 95% CI 2-sided [0 to 0.15]

2. Secondary Outcome: Change From Baseline in Morning Peak Expiratory Flow (PEF) (L/Min) at Home at Week 12
Description: The changes from baseline of weekly average of morning PEF (L/min) are compared between benralizumab 30 mg Q4W and placebo by using the mixed-effect model for repeated measures (MMRM) with baseline blood eosinophil count (≥300 cells/μL or <300 cells/μL), protocol specified visit, region (Europe or North America) and treatment*visit interaction as fixed effects and baseline morning PEF (L/min) as a covariate.
  Changes at Week 12 were calculated based on patients with both baseline and Week 12.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11 and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Benralizumab 30 mg Q4W | Placebo
Number analyzed (Participants) | 106 | 105
L/min
  Baseline | 307.413 (95.9467) | 308.226 (113.5895)
  Week 12 | 311.041 (101.8169) | 304.037 (113.2538)
  Change from baseline at Week 12 | 1.675 (56.5182) | -6.196 (45.3077)
Statistical Analysis 1: Comparison: Benralizumab 30 mg Q4W vs Placebo; Test type: Superiority or Other; p = 0.233, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Difference of Least Square Means = 8.84, 95% CI 2-sided [-5.74 to 23.42]

3. Secondary Outcome: Change From Baseline in Evening Peak Expiratory Flow (PEF) (L/Min) at Home at Week 12
Description: The changes from baseline of weekly average of evening PEF (L/min) are compared between benralizumab 30 mg Q4W and placebo by using the mixed-effect model for repeated measures (MMRM) with baseline blood eosinophil count (≥300 cells/μL or <300 cells/μL), protocol specified visit, region (Europe or North America) and treatment*visit interaction as fixed effects and baseline evening PEF (L/min) as a covariate.
  Changes at Week 12 were calculated based on patients with both baseline and Week 12.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11 and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Benralizumab 30 mg Q4W | Placebo
Number analyzed (Participants) | 106 | 105
L/min
  Baseline | 326.948 (97.4034) | 316.743 (116.6919)
  Week 12 | 330.719 (106.7579) | 316.047 (118.7000)
  Change from baseline at Week 12 | 1.361 (51.9979) | -2.956 (47.9136)
Statistical Analysis 1: Comparison: Benralizumab 30 mg Q4W vs Placebo; Test type: Superiority or Other; p = 0.456, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Difference of Least Square Means = 5.29, 95% CI 2-sided [-8.67 to 19.25]

4. Secondary Outcome: Change From Baseline in Total Asthma Symptom Score at Week 12
Description: Asthma symptoms were recorded by the patient each morning and evening in the asthma daily diary. Symptoms were recorded using a scale of 0-3, where 0 indicates no asthma symptoms. The daily asthma symptom total score was calculated by taking the sum of the daytime score recorded in the evening and the nighttime score recorded the following morning. The weekly total asthma score was averaged from the daily scores over a 7 day period, with score ranging from 0 to 6, where 0 indicates no asthma symptoms. The changes from baseline of weekly total asthma score are compared between benralizumab 30 mg Q4W and placebo by using the mixed-effect model repeated measures (MMRM) with baseline blood eosinophil count (≥300 cells/μL or <300 cells/μL), protocol specified visit, region (Europe or North America) and treatment*visit interaction as fixed effects and baseline total asthma score as a covariate.
  Changes at Week 12 were calculated based on patients with both baseline and Week 12.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11 and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg Q4W | Placebo
Number analyzed (Participants) | 106 | 105
Scores on a scale
  Baseline | 1.934 (0.9310) | 1.952 (1.0375)
  Week 12 | 1.326 (1.0448) | 1.541 (1.1208)
  Change from baseline at Week 12 | -0.567 (0.7875) | -0.420 (0.8767)
Statistical Analysis 1: Comparison: Benralizumab 30 mg Q4W vs Placebo; Test type: Superiority or Other; p = 0.266, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Difference of Least Square Means = -0.13, 95% CI 2-sided [-0.35 to 0.10]

5. Secondary Outcome: Change From Baseline in Total Asthma Rescue Medication Use (Puffs) at Week 12
Description: The number of rescue medication inhalations and nebulizer treatments taken were recorded by the patient in the asthma daily diary twice daily. The number of inhalations (puffs) per day was calculated as [number of night inhaler puffs] + 2 x [number of night nebulizer times] + number of day inhaler puffs + 2 x [number of day nebulizer times]. The changes from baseline in weekly total asthma rescue medication use (puffs) are compared between benralizumab 30 mg Q4W and placebo by using the mixed-effect model repeated measures (MMRM) with baseline blood eosinophil count (≥300 cells/μL or <300 cells/μL), protocol specified visit, region (Europe or North America) and treatment*visit interaction as fixed effects and baseline total asthma rescue medication use (puffs) as a covariate.
  Changes at Week 12 were calculated based on patients with both baseline and Week 12.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11 and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Puffs per day
Arm/Group | Benralizumab 30 mg Q4W | Placebo
Number analyzed (Participants) | 106 | 105
Puffs per day
  Baseline | 2.953 (3.0794) | 2.641 (3.0671)
  Week 12 | 1.647 (2.4782) | 2.070 (2.6848)
  Change from baseline at Week 12 | -1.098 (2.3588) | -0.665 (2.2744)
Statistical Analysis 1: Comparison: Benralizumab 30 mg Q4W vs Placebo; Test type: Superiority or Other; p = 0.200, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Difference of Least Square Means = -0.36, 95% CI 2-sided [-0.91 to 0.19]

6. Secondary Outcome: Change From Baseline in Proportion of Nights With Nocturnal Awakenings at Week 12
Description: Nocturnal awakenings due to asthma symptoms and requiring rescue medication use was recorded by the patient in the asthma daily diary each morning. Proportion of nights with nocturnal awakenings was defined as the number of nights with awakenings due to asthma and requiring rescue medication divided by number of nights with data for awakening due to asthma. The outcome variable for proportion of nights with nocturnal awakenings was the change from baseline at Week 12 in weekly proportion of nights with nocturnal awakenings. The changes are compared between benralizumab 30 mg Q4W and placebo by using the mixed-effect model repeated measures (MMRM) with baseline blood eosinophil count (≥300 cells/μL or <300 cells/μL), protocol specified visit, region (Europe or North America) and treatment*visit interaction as fixed effects and baseline proportion of nights with nocturnal awakenings as a covariate.
  Changes at Week 12 were calculated based on patients with both baseline and Week 12.
Time Frame: Baseline, Week 1, Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9, Week 10, Week 11 and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Proportion of nights
Arm/Group | Benralizumab 30 mg Q4W | Placebo
Number analyzed (Participants) | 106 | 105
Proportion of nights
  Baseline | 0.246 (0.2924) | 0.279 (0.3326)
  Week 12 | 0.086 (0.2003) | 0.144 (0.2796)
  Change from baseline at Week 12 | -0.158 (0.2515) | -0.139 (0.2659)
Statistical Analysis 1: Comparison: Benralizumab 30 mg Q4W vs Placebo; Test type: Superiority or Other; p = 0.380, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Difference of Least Square Means = -0.03, 95% CI 2-sided [-0.08 to 0.03]

7. Secondary Outcome: Change From Baseline in Mean ACQ-6 Score at Week 12
Description: The asthma control questionnaire, ACQ-6, consists of six questions; all assessed on a 7-point scale from 0 to 6, where 0 represents good control and 6 represents poor control. The overall score is the mean of the responses to each of the six questions. The changes from baseline of ACQ-6 score are compared between benralizumab 30 mg Q4W and placebo by using the mixed-effect repeated measures (MMRM) with baseline blood eosinophil count (≥300 cells/μL or <300 cells/μL), protocol specified visit (Week 4, Week 8, Week 12), region (Europe or North America) and treatment*visit interaction as fixed effects and baseline ACQ-6 score as a covariate.
  Changes at Week 12 were calculated based on patients with both baseline and Week 12.
Time Frame: Baseline, Week 4, Week 8 and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg Q4W | Placebo
Number analyzed (Participants) | 106 | 105
Scores on a scale
  Baseline | 2.119 (0.8423) | 2.092 (0.8975)
  Week 12 | 1.428 (0.8621) | 1.568 (1.0090)
  Change from baseline at Week 12 | -0.714 (0.8700) | -0.495 (0.7908)
Statistical Analysis 1: Comparison: Benralizumab 30 mg Q4W vs Placebo; Test type: Superiority or Other; p = 0.114, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Difference of Least Square Means = -0.17, 95% CI 2-sided [-0.39 to 0.04]

8. Secondary Outcome: Asthma Exacerbations
Description: An asthma exacerbation was defined as a worsening of asthma that led to use of systemic corticosteroids for at least 3 days (a single depo-injectable dose of corticosteroids was considered equivalent to a 3-day course of systemic corticosteroids) or an emergency room or urgent care visit (defined as evaluation and treatment for <24 hours in an emergency department or urgent care center) due to asthma that required systemic corticosteroids (as per above) or an inpatient hospitalization (defined as admission to an inpatient facility and/or evaluation and treatment in a healthcare facility for ≥24 hours) due to asthma. Number of patients experiencing an event included in the definition of asthma exacerbation was presented.
Time Frame: Up to Week 12
Population: as for outcome 1
Measure: Number; unit: Patients per number of exacerbations
Arm/Group | Benralizumab 30 mg Q4W | Placebo
Number analyzed (Participants) | 106 | 105
Patients per number of exacerbations
  0 exacerbation | 105 | 103
  1 exacerbation | 0 | 2
  2 exacerbations | 1 | 0

9. Secondary Outcome: Change From Baseline in AQLQ(S)+12 Total and Domain Scores at Week 12
Description: The asthma quality of life questionnaire for 12 years and older, AQLQ(S)+12, consists of 32 questions; all assessed on a 7-point scale from 7 to 1, where 7 represents no impairment and 1 represents severe impairment. The 4 individual domain scores (symptoms, activity limitations, emotional function, and environmental stimuli) are the means of the responses to the questions in each of the domains. The overall score is calculated as the mean response to all questions. The changes from baseline of AQLQ(S)+12 score are compared between benralizumab 30 mg Q4W and placebo by using the analyse of covariance (ANCOVA) with baseline blood eosinophil count (≥300 cells/μL or <300 cells/μL) and region (Europe or North America) as fixed effects and baseline AQLQ(S)+12 score as a covariate.
  Changes at Week 12 were calculated based on patients with both baseline and Week 12.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Benralizumab 30 mg Q4W | Placebo
Number analyzed (Participants) | 106 | 105
Scores on a scale
  Total score - Baseline | 4.825 (0.9787) | 4.895 (1.0339)
  Total score - W12 | 5.415 (0.9478) | 5.284 (1.0851)
  Total score - CFB at W12 | 0.585 (0.8675) | 0.357 (0.7979)
  Symptoms score - Baseline | 4.649 (1.0367) | 4.692 (1.0830)
  Symptoms score - W12 | 5.380 (1.0076) | 5.212 (1.1373)
  Symptoms score - CFB at W12 | 0.727 (0.9890) | 0.483 (0.9243)
  Activity limitations score - Baseline | 5.017 (1.0029) | 5.048 (1.0277)
  Activity limitations score - W12 | 5.503 (0.9672) | 5.343 (1.0803)
  Activity limitations score - CFB at W12 | 0.481 (0.8156) | 0.275 (0.8105)
  Emotional function score - Baseline | 4.95 (1.277) | 5.04 (1.373)
  Emotional function score - W12 | 5.54 (1.215) | 5.45 (1.307)
  Emotional function score - CFB at W12 | 0.57 (1.094) | 0.35 (1.014)
  Environmental stimuli score - Baseline | 4.658 (1.3320) | 4.905 (1.3554)
  Environmental stimuli score - W12 | 5.120 (1.2910) | 5.130 (1.3372)
  Environmental stimuli score - CFB at W12 | 0.466 (1.0135) | 0.216 (0.9505)
Statistical Analysis 1: Comparison: Benralizumab 30 mg Q4W vs Placebo; Parameter: Total score; Test type: Superiority or Other; p = 0.055, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Difference of Least Square Means = 0.21, 95% CI 2-sided [0 to 0.42]
Statistical Analysis 2: Comparison: Benralizumab 30 mg Q4W vs Placebo; Parameter: Symptoms score; Test type: Superiority or Other; p = 0.063, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Difference of Least Square Means = 0.23, 95% CI 2-sided [-0.01 to 0.47]
Statistical Analysis 3: Comparison: Benralizumab 30 mg Q4W vs Placebo; Parameter: Activity limitation score; Test type: Superiority or Other; p = 0.061, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Difference of Least Square Means = 0.20, 95% CI 2-sided [-0.01 to 0.41]
Statistical Analysis 4: Comparison: Benralizumab 30 mg Q4W vs Placebo; Parameter: Emotional function score; Test type: Superiority or Other; p = 0.156, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Difference of Least Square Means = 0.19, 95% CI 2-sided [-0.07 to 0.45]
Statistical Analysis 5: Comparison: Benralizumab 30 mg Q4W vs Placebo; Parameter: Environmental stimuli score; Test type: Superiority or Other; p = 0.135, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Difference of Least Square Means = 0.19, 95% CI 2-sided [-0.06 to 0.44]

10. Secondary Outcome: Serum Concentrations (ng/mL)
Description: Blood samples (processed to serum) for pharmacokinetic assessments were collected from all patients at baseline prior to first benralizumab administration at Day 1, at the Week 12 visit or the IP discontinuation visit, and at the Week 20 follow-up visit. Serum concentrations of benralizumab were determined using a validated electrochemiluminescent (ECL) immunoassay.
Time Frame: Baseline, Week 12 and Week 20
Population: The pharmacokinetic (PK) analysis set comprised all patients who received benralizumab and from whom PK blood samples were obtained are assumed not to be affected by factors such as protocol violations. Those patients who had at least 1 quantifiable serum PK observation post first dose were included in the PK analysis dataset.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Benralizumab 30 mg Q4W | Placebo
Number analyzed (Participants) | 103 | 0
ng/mL
  Pre- 1st dose | NA (NA) — All patients had concentration below the limit of quantification (3.86 ng/mL). |
  Week 12 | 999.16 (95.53) |
  Week 20 | 59.04 (317.71) |

11. Secondary Outcome: Peripheral Blood Eosinophil Levels
Description: Peripheral blood eosinophil levels assessments were collected from all patients at baseline prior to first benralizumab administration at Day 1, at the Week 12 visit or the IP discontinuation visit, and at the Week 20 follow-up visit.
  Changes at Week 12 (respectively at Week 20) were calculated based on patients with both baseline and Week 12 (respectively Week 20).
Time Frame: Baseline, Week 12 and Week 20
Population: The safety analysis set comprised all patients who received at least one dose of IP. Patients were classified according to the treatment they actually received. A patient who has on one or several occasions received active treatment was classified as active.
Measure: Median (Full Range); unit: Cells/µL
Arm/Group | Benralizumab 30 mg Q4W | Placebo
Number analyzed (Participants) | 106 | 105
Cells/µL
  Baseline | 170 [30 to 1060] | 220 [40 to 1140]
  Week 12 | 0.00 [0 to 110] | 230 [30 to 1000]
  Change from baseline at Week 12 | -170 [-1060 to 40] | 10 [-710 to 910]
  Week 20 | 0 [0 to 490] | 210 [40 to 1440]
  Change from Baseline at Week 20 | -160 [-1060 to 130] | 10 [-400 to 910]

ADVERSE EVENTS:
Time Frame: AEs, including SAEs, in the on-study period were defined as those with onset between day of the first dose of study treatment and last scheduled follow-up visit, inclusive, up to 20 weeks.
Description: The safety analysis set comprised all patients who received at least one dose of IP. Patients were classified according to the treatment they actually received. A patient who has on one or several occasions received active treatment was classified as active.
  No subject received wrong dose in the study.
Arm/Group | Benralizumab 30 mg Q4W | Placebo
Serious Adverse Events (participants affected / at risk) | 2/106 | 2/105
Other Adverse Events (participants affected / at risk) | 19/106 | 14/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab 30 mg Q4W (N=106) | Placebo (N=105)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Benralizumab 30 mg Q4W (N=106) | Placebo (N=105)
Nasopharyngitis (Infections and infestations) | 8 (8) | 8 (9)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 5 (5)
Headache (Nervous system disorders) | 4 (7) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
≥ 60 days prior to submission of material for publication/presentation, Institution and PI shall jointly provide AZ with material for review. No publication/presentation may include any of AZ's Confidential Information without AZ's written approval. AZ can request Inst. and PI to withhold material from submission for publication/presentation for an additional 90 days to allow AZ to establish and preserve its proprietary rights in the material being submitted for publication or presentation.